CLINICAL TRIAL: NCT01410604
Title: Inflammatory Mediators in Obese Adolescents With Insulin Resistance Following Metformin Treatment: Controlled Randomized Clinical Trial
Brief Title: Adipokines in Obese Adolescents With Insulin Resistance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Regional de Alta Especialidad del Bajio (Other)
Collaborators: Hospital Infantil de Mexico Federico Gomez (Other)
Responsible Party: Principal Investigator, Maria Lola Evia-Viscarra, Pediatrics Endocrinology, Hospital Regional de Alta Especialidad del Bajio
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 010-08
Record Dates: First submitted 2011-08-04; First posted 2011-08-05 (Estimated); Results first posted 2012-04-23 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Obesity
Keywords: Metformin; Obesity; Insulin resistance; Interleukin six; Adiponectin; High sensitivity C reactive protein.; Tumour Necrosis Factor alpha
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Experimental): Tablet of 500 mg metformin, oral every 12 hours (total metformin dose of 1 g/day) for 3 months.
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Tablet of 500 mg oral placebo every 12 hours for 3 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Tablet of 500 mg metformin, oral every 12 hours (total metformin dose of 1 g/day) for 3 months.
  Other Names: Dabex
  Arms: Metformin
Drug: Placebo — Tablet of 500 mg oral placebo every 12 hours for 3 months.
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare serum concentrations of inflammatory cytokines, interleukin 6 (IL-6), High-sensitivity C-reactive protein (hs-CRP), adiponectin, and tumour necrosis factor alpha (TNFα), before and after three months treatment with metformin in obese adolescents with insulin resistance (IR).

DETAILED DESCRIPTION:
The increased prevalence of obesity in pediatric patients is a public health problem particularly because of the difficulties involved with changing lifestyles. Current studies of obese children and adolescents show increased insulin resistance (IR) and chronic inflammatory states. These conditions increase the risk of disability and/or premature death.

The current treatment schemes for obese children are conservative and are focused on changing their lifestyles (exercise and dietary plans). However, metabolic conditions, such as IR, dyslipidemia, and inflammatory processes, are perpetuated.

Metformin is a biguanide that is used for adolescents with diabetes mellitus and polycystic ovarian syndrome. Several clinical trials with metformin for obese pediatric patients have observed decreases in IR, decreases in weight, and improvements in lipid metabolism.

Adipose tissue is not only an energy repository, but also plays an immunological role by the secretion of cytokines. Both overweight adults and adolescents show decreases in adiponectin levels and increases in tumor necrosis factor alpha (TNFα) and interleukin 6 (IL-6). IL-6 can stimulate the production of high-sensitivity C-reactive protein (hs-CRP), which is considered to be a risk marker for the development of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Obesity defined as Body Mass Index (BMI) ≥ percentile 95
* Tanner stage ≥ 2
* Insulin resistance defined as Basal insulin > 15 µU/mL or Homeostasis Model Assessment index (HOMA) > 4.5
* Patients' parents signed written consents when they and their adolescent children agreed to enroll

Exclusion Criteria:

* Glucose intolerance
* Diabetes mellitus (type 1 or 2)
* Anemia (Hb < 10 g/dL)
* Plasma creatinine > 1.4 mg/dL
* Abnormal hepatic function
* Any associated Disease (Pulmonary, Infection, Autoimmune Disease)
* History of lactic acidosis

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2007-01; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Evia-Viscarra, M.D., Principal Investigator — Hospital Regional de Alta Especialidad del Bajio; Edel R Rodea-Montero, Statistician, Study Chair — Hospital Regional de Alta Especialidad del Bajio; Evelia Apolinar-Jiménez, Nutrition, Study Chair — Hospital Regional de Alta Especialidad del Bajio; Leticia M García-Morales, M.D., Study Chair — Hospital Infantil de Mexico Federico Gomez; Constanza Leaños-Pérez, M.D., Study Chair — Hospital Infantil de Mexico Federico Gomez; Mireya Figueroa-Barrón, Chemestry, Study Chair — Hospital Infantil de Mexico Federico Gomez; Dolores Sánchez-Fierros, Chemestry, Study Chair — Hospital Infantil de Mexico Federico Gomez; Nathalie Muñoz-Noriega, Nutrition, Study Chair — Hospital Regional de Alta Especialidad del Bajio; Juan G Reyes-García, M.D., Study Chair — Escuela Superior de Medicina del IPN
Locations (2):
- Mexico (2):
  - Hospital Regional de Alta Especialidad del Bajío, León, Guanajuato
  - Hospital Infantil de México Federico Gómez, Mexico City, Mexico City

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). CDC grand rounds: childhood obesity in the United States. MMWR Morb Mortal Wkly Rep. 2011 Jan 21;60(2):42-6. PMID 21248681
- [Background] Wilfley DE, Tibbs TL, Van Buren DJ, Reach KP, Walker MS, Epstein LH. Lifestyle interventions in the treatment of childhood overweight: a meta-analytic review of randomized controlled trials. Health Psychol. 2007 Sep;26(5):521-32. doi: 10.1037/0278-6133.26.5.521. PMID 17845100
- [Background] Zeller M, Kirk S, Claytor R, Khoury P, Grieme J, Santangelo M, Daniels S. Predictors of attrition from a pediatric weight management program. J Pediatr. 2004 Apr;144(4):466-70. doi: 10.1016/j.jpeds.2003.12.031. PMID 15069394
- [Background] Ten S, Maclaren N. Insulin resistance syndrome in children. J Clin Endocrinol Metab. 2004 Jun;89(6):2526-39. doi: 10.1210/jc.2004-0276. PMID 15181020
- [Background] Chiarelli F, Marcovecchio ML. Insulin resistance and obesity in childhood. Eur J Endocrinol. 2008 Dec;159 Suppl 1:S67-74. doi: 10.1530/EJE-08-0245. Epub 2008 Sep 19. PMID 18805916
- [Background] Cruz ML, Weigensberg MJ, Huang TT, Ball G, Shaibi GQ, Goran MI. The metabolic syndrome in overweight Hispanic youth and the role of insulin sensitivity. J Clin Endocrinol Metab. 2004 Jan;89(1):108-13. doi: 10.1210/jc.2003-031188. PMID 14715836
- [Background] Visser M, Bouter LM, McQuillan GM, Wener MH, Harris TB. Low-grade systemic inflammation in overweight children. Pediatrics. 2001 Jan;107(1):E13. doi: 10.1542/peds.107.1.e13. PMID 11134477
- [Background] Freedman DS, Mei Z, Srinivasan SR, Berenson GS, Dietz WH. Cardiovascular risk factors and excess adiposity among overweight children and adolescents: the Bogalusa Heart Study. J Pediatr. 2007 Jan;150(1):12-17.e2. doi: 10.1016/j.jpeds.2006.08.042. PMID 17188605
- [Background] Beauloye V, Zech F, Tran HT, Clapuyt P, Maes M, Brichard SM. Determinants of early atherosclerosis in obese children and adolescents. J Clin Endocrinol Metab. 2007 Aug;92(8):3025-32. doi: 10.1210/jc.2007-0619. Epub 2007 May 22. PMID 17519311
- [Background] Berenson GS, Srinivasan SR, Bao W, Newman WP 3rd, Tracy RE, Wattigney WA. Association between multiple cardiovascular risk factors and atherosclerosis in children and young adults. The Bogalusa Heart Study. N Engl J Med. 1998 Jun 4;338(23):1650-6. doi: 10.1056/NEJM199806043382302. PMID 9614255
- [Background] Type 2 diabetes in children and adolescents. American Diabetes Association. Pediatrics. 2000 Mar;105(3 Pt 1):671-80. doi: 10.1542/peds.105.3.671. No abstract available. PMID 10699131
- [Background] SEARCH for Diabetes in Youth Study Group; Liese AD, D'Agostino RB Jr, Hamman RF, Kilgo PD, Lawrence JM, Liu LL, Loots B, Linder B, Marcovina S, Rodriguez B, Standiford D, Williams DE. The burden of diabetes mellitus among US youth: prevalence estimates from the SEARCH for Diabetes in Youth Study. Pediatrics. 2006 Oct;118(4):1510-8. doi: 10.1542/peds.2006-0690. PMID 17015542
- [Background] Kay JP, Alemzadeh R, Langley G, D'Angelo L, Smith P, Holshouser S. Beneficial effects of metformin in normoglycemic morbidly obese adolescents. Metabolism. 2001 Dec;50(12):1457-61. doi: 10.1053/meta.2001.28078. PMID 11735093
- [Background] Love-Osborne K, Sheeder J, Zeitler P. Addition of metformin to a lifestyle modification program in adolescents with insulin resistance. J Pediatr. 2008 Jun;152(6):817-22. doi: 10.1016/j.jpeds.2008.01.018. Epub 2008 Mar 19. PMID 18492523
- [Background] Srinivasan S, Ambler GR, Baur LA, Garnett SP, Tepsa M, Yap F, Ward GM, Cowell CT. Randomized, controlled trial of metformin for obesity and insulin resistance in children and adolescents: improvement in body composition and fasting insulin. J Clin Endocrinol Metab. 2006 Jun;91(6):2074-80. doi: 10.1210/jc.2006-0241. Epub 2006 Apr 4. PMID 16595599
- [Background] Trayhurn P, Beattie JH. Physiological role of adipose tissue: white adipose tissue as an endocrine and secretory organ. Proc Nutr Soc. 2001 Aug;60(3):329-39. doi: 10.1079/pns200194. PMID 11681807
- [Background] Stefan N, Bunt JC, Salbe AD, Funahashi T, Matsuzawa Y, Tataranni PA. Plasma adiponectin concentrations in children: relationships with obesity and insulinemia. J Clin Endocrinol Metab. 2002 Oct;87(10):4652-6. doi: 10.1210/jc.2002-020694. PMID 12364452
- [Background] Weiss R, Dufour S, Groszmann A, Petersen K, Dziura J, Taksali SE, Shulman G, Caprio S. Low adiponectin levels in adolescent obesity: a marker of increased intramyocellular lipid accumulation. J Clin Endocrinol Metab. 2003 May;88(5):2014-8. doi: 10.1210/jc.2002-021711. PMID 12727947
- [Background] Moon YS, Kim DH, Song DK. Serum tumor necrosis factor-alpha levels and components of the metabolic syndrome in obese adolescents. Metabolism. 2004 Jul;53(7):863-7. doi: 10.1016/j.metabol.2004.02.007. PMID 15254878
- [Background] Herder C, Schneitler S, Rathmann W, Haastert B, Schneitler H, Winkler H, Bredahl R, Hahnloser E, Martin S. Low-grade inflammation, obesity, and insulin resistance in adolescents. J Clin Endocrinol Metab. 2007 Dec;92(12):4569-74. doi: 10.1210/jc.2007-0955. Epub 2007 Oct 2. PMID 17911172
- [Background] Cartier A, Lemieux I, Almeras N, Tremblay A, Bergeron J, Despres JP. Visceral obesity and plasma glucose-insulin homeostasis: contributions of interleukin-6 and tumor necrosis factor-alpha in men. J Clin Endocrinol Metab. 2008 May;93(5):1931-8. doi: 10.1210/jc.2007-2191. Epub 2008 Mar 4. PMID 18319319
- [Background] Ford ES, Galuska DA, Gillespie C, Will JC, Giles WH, Dietz WH. C-reactive protein and body mass index in children: findings from the Third National Health and Nutrition Examination Survey, 1988-1994. J Pediatr. 2001 Apr;138(4):486-92. doi: 10.1067/mpd.2001.112898. PMID 11295710
- [Background] Hiura M, Kikuchi T, Nagasaki K, Uchiyama M. Elevation of serum C-reactive protein levels is associated with obesity in boys. Hypertens Res. 2003 Jul;26(7):541-6. doi: 10.1291/hypres.26.541. PMID 12924621
- [Background] Freedman DS, Sherry B. The validity of BMI as an indicator of body fatness and risk among children. Pediatrics. 2009 Sep;124 Suppl 1:S23-34. doi: 10.1542/peds.2008-3586E. PMID 19720664
- [Background] Cole TJ, Bellizzi MC, Flegal KM, Dietz WH. Establishing a standard definition for child overweight and obesity worldwide: international survey. BMJ. 2000 May 6;320(7244):1240-3. doi: 10.1136/bmj.320.7244.1240. PMID 10797032
- [Background] Kuczmarski RJ, Ogden CL, Guo SS, Grummer-Strawn LM, Flegal KM, Mei Z, Wei R, Curtin LR, Roche AF, Johnson CL. 2000 CDC Growth Charts for the United States: methods and development. Vital Health Stat 11. 2002 May;(246):1-190. PMID 12043359
- [Background] Reaven GM, Chen YD, Hollenbeck CB, Sheu WH, Ostrega D, Polonsky KS. Plasma insulin, C-peptide, and proinsulin concentrations in obese and nonobese individuals with varying degrees of glucose tolerance. J Clin Endocrinol Metab. 1993 Jan;76(1):44-8. doi: 10.1210/jcem.76.1.8421101.
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Keskin M, Kurtoglu S, Kendirci M, Atabek ME, Yazici C. Homeostasis model assessment is more reliable than the fasting glucose/insulin ratio and quantitative insulin sensitivity check index for assessing insulin resistance among obese children and adolescents. Pediatrics. 2005 Apr;115(4):e500-3. doi: 10.1542/peds.2004-1921. Epub 2005 Mar 1. PMID 15741351
- [Background] Weyer C, Funahashi T, Tanaka S, Hotta K, Matsuzawa Y, Pratley RE, Tataranni PA. Hypoadiponectinemia in obesity and type 2 diabetes: close association with insulin resistance and hyperinsulinemia. J Clin Endocrinol Metab. 2001 May;86(5):1930-5. doi: 10.1210/jcem.86.5.7463. PMID 11344187
- [Background] Fruebis J, Tsao TS, Javorschi S, Ebbets-Reed D, Erickson MR, Yen FT, Bihain BE, Lodish HF. Proteolytic cleavage product of 30-kDa adipocyte complement-related protein increases fatty acid oxidation in muscle and causes weight loss in mice. Proc Natl Acad Sci U S A. 2001 Feb 13;98(4):2005-10. doi: 10.1073/pnas.98.4.2005. Epub 2001 Feb 6. PMID 11172066
- [Background] Perea-Martinez A, Carbajal R.L, Rodriguez H.R, Zarco R.J, Barrios F.R, Loredo A.A, et al. Association of comorbidity with obesity in mexican children and adolescents. Pediatrics 2008;121(2):S149-S150
- [Background] Yeh ET. High-sensitivity C-reactive protein as a risk assessment tool for cardiovascular disease. Clin Cardiol. 2005 Sep;28(9):408-12. doi: 10.1002/clc.4960280905. PMID 16250263
- [Background] Balagopal P, George D, Patton N, Yarandi H, Roberts WL, Bayne E, Gidding S. Lifestyle-only intervention attenuates the inflammatory state associated with obesity: a randomized controlled study in adolescents. J Pediatr. 2005 Mar;146(3):342-8. doi: 10.1016/j.jpeds.2004.11.033. PMID 15756217
- [Background] Monzillo LU, Hamdy O, Horton ES, Ledbury S, Mullooly C, Jarema C, Porter S, Ovalle K, Moussa A, Mantzoros CS. Effect of lifestyle modification on adipokine levels in obese subjects with insulin resistance. Obes Res. 2003 Sep;11(9):1048-54. doi: 10.1038/oby.2003.144. PMID 12972674
- [Background] Huang NL, Chiang SH, Hsueh CH, Liang YJ, Chen YJ, Lai LP. Metformin inhibits TNF-alpha-induced IkappaB kinase phosphorylation, IkappaB-alpha degradation and IL-6 production in endothelial cells through PI3K-dependent AMPK phosphorylation. Int J Cardiol. 2009 May 15;134(2):169-75. doi: 10.1016/j.ijcard.2008.04.010. Epub 2008 Jul 1. PMID 18597869
- [Background] Zhou G, Myers R, Li Y, Chen Y, Shen X, Fenyk-Melody J, Wu M, Ventre J, Doebber T, Fujii N, Musi N, Hirshman MF, Goodyear LJ, Moller DE. Role of AMP-activated protein kinase in mechanism of metformin action. J Clin Invest. 2001 Oct;108(8):1167-74. doi: 10.1172/JCI13505. PMID 11602624
- [Derived] Evia-Viscarra ML, Rodea-Montero ER, Apolinar-Jimenez E, Munoz-Noriega N, Garcia-Morales LM, Leanos-Perez C, Figueroa-Barron M, Sanchez-Fierros D, Reyes-Garcia JG. The effects of metformin on inflammatory mediators in obese adolescents with insulin resistance: controlled randomized clinical trial. J Pediatr Endocrinol Metab. 2012;25(1-2):41-9. doi: 10.1515/jpem-2011-0469. PMID 22570949

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled between January 2007 and December 2009 in the Pediatric Obesity Clinics (POC) from third level Mexican Hospitals: the HMFG, located in the Federal District (country's capital), and the HRAEB, located in the city of Leon in the state of Guanajauto.
Period: Overall Study
Arm/Group | Metformin | Placebo
Started | 15 | 16
Completed | 12 | 14
Not Completed | 3 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 16 | 31
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 12.56 (2.25) | 14.12 (1.20) | 13.37 (1.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  Mexico | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Adiponectin
Description: Change from baseline in Adiponectin after 3 months of treatment.
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 12 | 14
µg/mL | -0.71 (4.29) | -7.52 (6.28)

2. Primary Outcome: High-sensitivity C-reactive Protein
Description: Change from baseline in High-sensitivity C-reactive protein after 3 months of treatment.
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 12 | 14
mg/dL | -1.26 (4.40) | -1.35 (13.60)

3. Primary Outcome: Interleukin 6
Description: Change from baseline in Interleukin 6 after 3 months of treatment.
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 12 | 14
pg/mL | -34.09 (145.72) | 16.42 (60.50)

4. Primary Outcome: Tumour Necrosis Factor Alpha
Description: Change from baseline in Tumour necrosis factor alpha after 3 months of treatment.
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 12 | 14
pg/mL | -34.08 (77.58) | -4.01 (31.82)

5. Secondary Outcome: Fasting Plasma Glucose
Description: Change from baseline in Fasting plasma glucose after 3 months of treatment.
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 12 | 14
mg/dL | -1.08 (11.39) | 1.71 (15.61)

6. Secondary Outcome: Fasting Insulin
Description: Change from baseline in Fasting insulin after 3 months of treatment.
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: µU/mL
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 12 | 14
µU/mL | -3.97 (23.28) | 11.03 (14.37)

7. Secondary Outcome: Body Mass Index
Description: Change from baseline in Body Mass Index after 3 months of treatment.
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 12 | 14
kg/m^2 | -0.74 (0.83) | -0.71 (0.85)

8. Secondary Outcome: Waist Circumference
Description: Change from baseline in Waist circumference after 3 months of treatment.
Time Frame: baseline and 3 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 12 | 14
cm | -0.57 (4.28) | -3.29 (5.24)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Metformin | Placebo
Serious Adverse Events (participants affected / at risk) | 2/15 | 1/16
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=15) | Placebo (N=16)
Epigastric pain (Gastrointestinal disorders) | 2 (2) | 1 (1) — Adverse effect characterized by " burning " epigastric pain

LIMITATIONS AND CAVEATS:
During the recruitment phase, 83 children who were diagnosed with obesity and acanthosis nigricans were evaluated. Of these, 45 did not have the insulin concentration values (>15 µU/mL) required to biochemically define Insulin Resistance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes